CLINICAL TRIAL: NCT00723866
Title: Combined Botulinum Toxin Type A With Modified Constraint-Induced Movement Therapy for Chronic Stroke Patients With Upper Extremity Spasticity
Brief Title: Botulinum Toxin Type A and Modified Constraint-Induced Movement Therapy for Poststroke Upper Extremity Spasticity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Kaohsiung Veterans General Hospital, Kaohsiung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VGHKS94-087
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2008-08-01 (Estimated); Status verified 2008-07

CONDITIONS: Stroke
Keywords: Botulinum toxin, Spasticity, Stroke, Rehabilitation.
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): BtxA+mCIMT (combination group)
  Interventions: Other: BtxA+mCIMT
- 2 (Placebo Comparator): BtxA+ conventional rehabilitation (control group)
  Interventions: Other: BtxA+ conventional rehabilitation

INTERVENTIONS:
Other: BtxA+mCIMT — The combination group receive BtxA+mCIMT for 2 hours/day, 3 days/week for 3 months.
  Other Names: the combination group
  Arms: 1
Other: BtxA+ conventional rehabilitation — The control group received for 2 hours/day, 3 days/week for 3 months.
  Other Names: the control group
  Arms: 2

SUMMARY:
Botulinum toxin type A (BtxA) injection and modified constraint-induced movement therapy (mCIMT) are both promising approaches to enhance recovery after stroke. However, the combined application of the two modalities has rarely been studied. The aim was to investigate whether combined BtxA and mCIMT would produce greater improvements in spasticity and upper extremity function than BtxA plus conventional rehabilitation in chronic stroke patients with upper extremity spasticity.

DETAILED DESCRIPTION:
Botulinum toxin type A (BtxA) injection and modified constraint-induced movement therapy (mCIMT)are both promising approaches to enhance recovery after stroke. However, the combined application of the two modalities has rarely been studied. To date, only a single case report addressed this issue. Theoretically, application of a mCIMT program with intensive functional tasks practice after spasticity reduction by BtxA may improve affected upper extremity function in patients with poststroke spasticity. The aim was to investigate whether combined BtxA and mCIMT would produce greater improvements in spasticity and upper extremity function than BtxA plus conventional rehabilitation in chronic stroke patients with upper extremity spasticity.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 80 years
* at least 1 year after a unilateral stroke
* modified ashworth scale (MAS) score > 3 in the elbow, wrist or finger flexors
* ability to actively extend > 10 degrees at metacarpophalangeal and interphalangeal joints and 20 degrees at wrist of the affected upper limb (minimal motor criteria).

Exclusion Criteria:

* presence of fixed joint contractures
* serious balance problems
* preexisting neurological deficits, neuromuscular diseases or uncontrolled medical conditions
* significant cognitive deficits (Mini-Mental Status Examination score < 24)
* excessive pain in the affected upper limb
* previous treatment with Botulinum toxin A, neurolytic agents or surgery for spasticity

All patients were not currently participating in any experimental studies and did not receive concomitant oral anti-spastic medication during the study period

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-12; Primary Completion 2007-11 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome assessed spasticity on the Modified Ashworth Scale. | MAS evaluated before BtxA injection, at 4 weeks, 3 months and 6 months postinjection.

SECONDARY OUTCOMES:
Secondary outcomes assessed real-world arm function (Motor Activity Log), laboratory motor activity (Action Research Arm Test) and patients' global satisfaction. | evaluated before BtxA injection, at 4 weeks, 3 months and 6 months postinjection.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Fen Sun, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation

REFERENCES:
- [Background] Sun SF, Hsu CW, Hwang CW, Hsu PT, Wang JL, Yang CL. Application of combined botulinum toxin type A and modified constraint-induced movement therapy for an individual with chronic upper-extremity spasticity after stroke. Phys Ther. 2006 Oct;86(10):1387-97. doi: 10.2522/ptj.20050262. PMID 17012643